CLINICAL TRIAL: NCT05266781
Title: A PROpensity Score Matching Analysis on ENDovascular vs Open Thoraco-Abdominal Aortic Aneurysm Repair . A Single-center, Retrospective-prospective, Observational Study/ EUnetHTA Core Model
Brief Title: A PROpensity Score Matching Analysis on ENDovascular vs Open Thoraco-Abdominal Aortic Aneurysm Repair (PRO-ENDO TAAA Study)
Acronym: PRO-ENDO TAAA
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Bertoglio Luca, Prof, IRCCS San Raffaele
Other Study IDs: PRO-ENDO TAAA study
Record Dates: First submitted 2022-02-23; First posted 2022-03-04 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Thoracoabdominal Aortic Aneurysms
MeSH Terms: conditions — Aortic Aneurysm, Thoracoabdominal | interventions — Wound Healing; Endovascular Aneurysm Repair

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Open surgical repair: Aneurysmectomy and aortic reconstruction with a surgical graft
  Interventions: Procedure: Surgical repair
- Endovascular repair: Off-the-shelf or custom-made Fenestrated/Branched-Endovascular Aortic Repair - F/BEVAR
  Interventions: Procedure: Endovascular repair

INTERVENTIONS:
Procedure: Surgical repair — Patients affected by a thoracoabdominal aortic aneurysm who received an open surgical repair (aneurysmectomy and aortic reconstruction with a surgical graft
  Groups: Open surgical repair
Procedure: Endovascular repair — Patients affected by a thoracoabdominal aortic aneurysm who received endovascular repair (with off-the-shelf or custom-made Fenestrated/Branched-Endovascular Aortic Repair - F/BEVAR)
  Groups: Endovascular repair

SUMMARY:
The purpose of the registry is to compare the surgical and endovascular approaches to the treatment of thoracoabdominal aortic aneurysms.

DETAILED DESCRIPTION:
The purpose of the study is to compare the surgical and endovascular approaches to the treatment of thoracoabdominal aortic aneurysms. In particular, the study aims at comparing the short- and mid-term mortality, morbidity and reintervention rate after open surgery or endovascular repair of thoracoabdominal aortic aneurysms in comparable cohorts of patients according to preoperative characteristics and evaluating the cost-effectiveness of both techniques, according to the EUnetHTA core model.

The study results will contribute to the creation of a HTA Report regarding endovascular technology to treat thoracoabdominal aortic aneurysms which will be evaluated by the appropriate Health Authorities.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by a thoracoabdominal aortic aneurysm who received an open surgical repair (aneurysmectomy and aortic reconstruction with a surgical graft) or endovascular repair (with off-the-shelf or custom-made Fenestrated/Branched-Endovascular Aortic Repair - F/BEVAR) between January 2013 and June 2021 at San Raffaele Hospital (Vascular Surgery Unit)
* Adult patients ≥18 years
* The patient is able to understand and sign the informed consent approved by the Ethics Committee of the San Raffaele Hospital

Exclusion Criteria:

* Patients treated with a hybrid approach (open surgical retrograde revascularization of renovisceral arteries followed by aneurysm exclusion with endograft)
* Patients treated with other endovascular techniques besides fenestrated or branched technology (e.g., physician-modified endografts, parallel grafts).
* Patients with a juxtarenal or pararenal aortic aneurysm
* Patients treated with F/BEVAR for a visceral artery patch aneurysm after open thoracoabdominal repair

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: We aim to include at least 650 patients in a 3-month period. Follow-up data will be recorded up to 1 year postoperatively. Data verification and analysis will request 2 months after study completion. The overall duration of the study will be 6 months
Sampling Method: Non-Probability Sample
Enrollment: 650 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
free survival | 1 year
  1 year aortic-related and all cause mortality
aortic-related reintervention | 1 year
  1 year clinical success

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crawford ES, Crawford JL, Safi HJ, Coselli JS, Hess KR, Brooks B, Norton HJ, Glaeser DH. Thoracoabdominal aortic aneurysms: preoperative and intraoperative factors determining immediate and long-term results of operations in 605 patients. J Vasc Surg. 1986 Mar;3(3):389-404. doi: 10.1067/mva.1986.avs0030389. PMID 3951025
- [Background] Bertoglio L, Grandi A, Melloni A, Kahlberg A, Melissano G, Chiesa R. Percutaneous AXillary Artery (PAXA) Access at the First Segment During Fenestrated and Branched Endovascular Aortic Procedures. Eur J Vasc Endovasc Surg. 2020 Jun;59(6):929-938. doi: 10.1016/j.ejvs.2020.01.027. Epub 2020 Feb 20. PMID 32089506
- [Background] Rocha RV, Lindsay TF, Friedrich JO, Shan S, Sinha S, Yanagawa B, Al-Omran M, Forbes TL, Ouzounian M. Systematic review of contemporary outcomes of endovascular and open thoracoabdominal aortic aneurysm repair. J Vasc Surg. 2020 Apr;71(4):1396-1412.e12. doi: 10.1016/j.jvs.2019.06.216. Epub 2019 Nov 2. PMID 31690525
- [Background] Rocha RV, Friedrich JO, Elbatarny M, Yanagawa B, Al-Omran M, Forbes TL, Lindsay TF, Ouzounian M. A systematic review and meta-analysis of early outcomes after endovascular versus open repair of thoracoabdominal aortic aneurysms. J Vasc Surg. 2018 Dec;68(6):1936-1945.e5. doi: 10.1016/j.jvs.2018.08.147. PMID 30470373